CLINICAL TRIAL: NCT02158936
Title: A Randomized, Double-blind, Placebo-controlled, Phase III, Multi-centre Study of Eltrombopag or Placebo in Combination With Azacitidine in Subjects With IPSS Intermediate-1, Intermediate 2 and High-risk Myelodysplastic Syndromes (MDS) SUPPORT: A StUdy of eltromboPag in myelodysPlastic SyndrOmes Receiving azaciTidine
Brief Title: A Study of Eltrombopag or Placebo in Combination With Azacitidine in Subjects With International Prognostic Scoring System (IPSS) Intermediate-1, Intermediate-2 or High-risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112121
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-09

CONDITIONS: Thrombocytopaenia
Keywords: thrombocytopenia; myelodysplastic syndromes; MDS; thrombopoietin; azacitidine; Eltrombopag; myelodysplastic syndromes (MDS)
MeSH Terms: conditions — Thrombocytopenia; Myelodysplastic Syndromes; Jacobs syndrome | interventions — eltrombopag; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Experimental): Eligible subject will receive a starting dose of eltrombopag of 200 milligrams (mg) (100 mg for subjects of East Asian heritage). Dose modifications of eltrombopag will be permitted by 100 mg increments (50 mg increments for East Asians) to a lowest dose of 100 mg (50 mg for East Asian heritage) or a maximum dose of 300 mg (150 mg for East Asian heritage) in order to maintain platelet counts at a safe and effective level (i.e. a level sufficient to avoid platelet transfusions and bleeding events). Subjects will receive azacitidine 75 mg/meter^2 subcutaneously once daily for 7 days (+/- 3 day treatment window permitted) every 28 days, for at least 6 cycles if tolerated and until they are no longer receiving benefit (defined as at least stable disease per the investigator's assessment) or until disease progression, death, or unacceptable toxicity/adverse event. The subject may receive eltrombopag daily for the full 28 days each cycle for as long as the subject is receiving azacitidine
  Interventions: Drug: Eltrombopag; Drug: Azacitidine
- Placebo (Placebo Comparator): Eligible subject will receive eltrombopag matching placebo. Subjects will receive azacitidine 75 mg/meter^2 subcutaneously once daily for 7 days (+/- 3 day treatment window permitted) every 28 days, for at least 6 cycles if tolerated and until they are no longer receiving benefit (defined as at least stable disease per the investigator's assessment) or until disease progression, death, or unacceptable toxicity/adverse event. The subject may receive eltrombopag daily for the full 28 days each cycle for as long as the subject is receiving azacitidine
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be round film-coated tablets containing eltrombopag equivalent to 50 mg (white to off-white), 200 mg and 300 mg (green) of eltrombopag free acid
  Arms: Eltrombopag
Drug: Azacitidine — Subcutaneous Injection (IV if local standard)
Drug: Placebo — Eltrombopag matching placebo tablets
  Arms: Placebo
Drug: Placebo — Eltrombopag matching placebo tablets will be supplied
  Arms: Placebo

SUMMARY:
Eltrombopag olamine (SB-497115-GR) is an orally bioavailable, small molecule thrombopoietin receptor agonist that may be beneficial in medical disorders associated with thrombocytopenia. Eltrombopag has been shown to increase platelet counts in patients with thrombocytopenia from various etiologies (Idiopathic thrombocytopenic purpura [ITP], liver disease, aplastic anemia and chemotherapy induced thrombocytopenia). Approximately 350 subjects will be randomized in a 1:1 ratio (175 into the eltrombopag arm and 175 into the placebo arm). Approximately 55 subjects will be enrolled into the azacitidine. Subjects with intermediate-1, intermediate-2 or high risk MDS by IPSS, and baseline platelet count of <75 Giga (10^9) per liter (Gi/L) will only be enrolled. This is a randomized, double-blind, parallel group, placebo-controlled study designed to explore the platelet supportive care effects of eltrombopag versus placebo in combination with the standard of care hypomethylating agent, azacitidine. The primary objective of this study is to determine the effect of eltrombopag versus placebo on the proportion of subjects who are platelet transfusion free during the first 4 cycles of azacitidine therapy. Key secondary endpoints include overall survival, disease response, and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years (For subjects in Taiwan, Age >= 20 years)
* MDS by World Health Organization (WHO) or French-American-British (FAB) classification
* Intermediate 1, intermediate 2 or high risk MDS by IPSS
* At least one platelet count < 75 Gi/L
* Eastern Cooperative Oncology Group (ECOG) Status 0-2
* Adequate baseline organ function defined by the criteria below: total bilirubin =< 1.5x the upper limit of normal (ULN) except for Gilbert's syndrome or cases clearly not indicative of inadequate liver function (i.e. elevation of indirect [haemolytic] bilirubin in the absence of alanine aminotransferase [ALT] abnormality); ALT =< 2.5xULN; creatinine =< 2.5xULN
* Subjects with a corrected QT interval (QTc) <450 milliseconds (msec) or <480msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), machine or manual overread. For subject eligibility and withdrawal, QTcF will be used. For purposes of data analysis, QTcF will be used. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period
* Subject is able to understand and comply with protocol requirements and instructions
* Subject has signed and dated informed consent
* Women must be either of non-child bearing potential, or women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception during the study and for 3 months following the last dose of study treatment
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of randomization until 16 weeks after the last dose of study treatment
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Previous treatment with hypomethylating agent or induction chemotherapy for MDS
* Proliferative type chronic myelomonocytic leukemia with white blood cell count >12 Gi/L at any time during the 28 days before Day 1
* History of treatment with eltrombopag, romiplostim or other thrombopoietin receptor (TPO-R) agonists
* Previous allogeneic stem-cell transplantation
* Known thrombophilic risk factors. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of investigational product (eltrombopag/placebo)
* Active and uncontrolled infections, including hepatitis B or C
* Human Immunodeficiency Virus (HIV) infection
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag or its excipient, or azacitidine, that contraindicates the subjects' participation
* Pregnant or lactating female
* Any serious and/or unstable pre-existing medical condition (including any advanced malignancy other than the disease under study), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (130):
- United States (10):
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Santa Fe
- Australia (5):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (7):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Steyr
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Lodelinsart
  - Novartis Investigative Site, Turnhout
- Brazil (7):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Sao Paulo - SP
- Canada (5):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Québec
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Koebenhavn Oe
- France (5):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pringy
- Germany (6):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (4):
  - Novartis Investigative Site, Chai Wan
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Shatin, New Territories
  - Novartis Investigative Site, Tuenmen
- Hungary (2):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
- Ireland (5):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, James Street
  - Novartis Investigative Site, Limerick
  - Novartis Investigative Site, Tallaght, Dublin
- Israel (6):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Reggio Calabria, Calabria
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Florence, Tuscany
- Mexico (2):
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Oaxaca City
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Novartis Investigative Site, Lima, Peru
- Poland (6):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Legnica
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Torun
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (5):
  - Novartis Investigative Site, Kaluga
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- Novartis Investigative Site, Seoul, South Korea
- Spain (14):
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, La Laguna (Santa Cruz de Tenerife)
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Majadahonda (Madrid)
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Oviedo
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pozuelo de Alarcon/Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón/Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Samsun

REFERENCES:
- [Derived] Dickinson M, Cherif H, Fenaux P, Mittelman M, Verma A, Portella MSO, Burgess P, Ramos PM, Choi J, Platzbecker U; SUPPORT study investigators. Azacitidine with or without eltrombopag for first-line treatment of intermediate- or high-risk MDS with thrombocytopenia. Blood. 2018 Dec 20;132(25):2629-2638. doi: 10.1182/blood-2018-06-855221. Epub 2018 Oct 10. PMID 30305280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 356 patients were enrolled in the study and 2 patients did not receive treatment.
Groups:
- Eltrombopag: Starting dose is 200 mg (100 mg for East Asian heritage). Dose modifications permitted by 100 mg increments (50 mg increments for East Asians) to a lowest dose of 100 mg (50 mg for East Asian heritage) or a maximum dose of 300 mg (150 mg for East Asian heritage) in order to maintain platelet counts at safe, effective level (level sufficient to avoid platelet transfusions and bleeding events). Subjects will receive Azacitidine 75 mg/meter^2 is administered subcutaneously once daily for 7 days every 28 days, for at least 6 cycles, if tolerated, until they are no longer receiving benefit (at least stable disease), disease progression, death, or unacceptable toxicity/adverse event. The subject may receive eltrombopag daily for the full 28 days each cycle if subject is receiving azacitidine
- Placebo: Subject will receive eltrombopag matching placebo. Subjects will receive azacitidine 75 mg/meter^2 subcutaneously once daily for 7 days (+/- 3 day treatment window permitted) every 28 days, for at least 6 cycles if tolerated and until they are no longer receiving benefit (defined as at least stable disease per the investigator's assessment) or until disease progression, death, or unacceptable toxicity/adverse event. The subject may receive matching placebo daily for the full 28 days each cycle for as long as the subject is receiving azacitidine
Period: Overall Study
Arm/Group | Eltrombopag | Placebo
Started | 179 | 177
Treated | 177 | 177
Untreated | 2 | 0
Completed | 0 | 0
Not Completed | 179 | 177
Not completed — Study closed/ terminated | 57 | 77
Not completed — Azacitidine tx discontinued | 53 | 46
Not completed — Adverse Event | 39 | 24
Not completed — Withdrawal by Subject | 15 | 16
Not completed — Physician Decision | 15 | 13
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag | Placebo | Total
Number analyzed (Participants) | 179 | 177 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (12.82) | 69.4 (10.58) | 68.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 53 | 122
  Male | 110 | 124 | 234
Race/Ethnicity, Customized [Number; unit: participants]
  White | 146 | 148 | 294
  East Asian/Japanese/S.E. Asian | 26 | 23 | 49
  Central/South Asian | 0 | 2 | 2
  Other | 4 | 4 | 8
  Missing | 3 | 0 | 3
IPSS risk score [Number; unit: participants] — A bone marrow examination for the determination of IPSS was performed during the screening period, or within 3 months prior to randomization. Assessment of bone marrow blasts was to be completed by bone marrow slide review. The patient's IPSS risk category is determined by adding together all of the IPSS scores within the three disease factors (blast cells, chromosomal changes, presence of cytopenias). That number is matched to one of the following four IPSS risk categories: Low, Intermediate-1, Intermediate-2, or High. The higher the score the higher the risk.
  participants
    Int - 1 (0.5-1.0) | 64 | 61 | 125
    Int - 2 (1.5 - 2.0) | 77 | 83 | 160
    High Risk (≥ 2.5) | 38 | 33 | 71
Platelet Count [Number; unit: participants]
  < 10 | 10 | 10 | 20
  ≥ 10 - <20 | 35 | 30 | 65
  ≥ 20 - <50 | 83 | 84 | 167
  ≥ 50 - <100 | 49 | 53 | 102
  ≥ 100 | 0 | 0 | 0
  missing | 2 | 0 | 2
Platelet transfusion dependence [Number; unit: participants]
  Yes | 29 | 37 | 66
  No | 150 | 140 | 290

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Platelet Transfusion Independent During Cycles 1-4 of Azacitidine Therapy
Description: A subject is defined as being platelet transfusion independent if they received no platelet transfusions within the first 4 cycles of treatment with azacitidine. Subjects who died or withdrew from investigational product within the first four cycles were treated as failures (i.e. not transfusion independent) in the analysis
Time Frame: 4 cycles (Cycle = 28 days)
Population: Intent-to-Treat population, comprised of all randomized patients
Measure: Number; unit: Participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
Participants
  Yes - platelet transfusion independent | 28 | 55
  No - platelet transfusion independent | 151 | 122
Statistical Analysis 1: Comparison: Eltrombopag vs Placebo; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — One sided p value; Stratified by Interactive Voice Response System (IVRS) stratification factors; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.21 to 0.65]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death due to any cause and deaths have been presented. Subjects still alive at the time of the analysis and subjects who have withdrawn from the study will be censored at the time of last contact
Time Frame: Randomization until death or end of study, approximately 2 years
Measure: Number; unit: deaths (events)
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
deaths (events) | 57 | 51
Statistical Analysis 1: Comparison: Eltrombopag vs Placebo; Confidence Intervals estimated using the Brookmeyer-Crowley method. Hazard ratios are estimated using the Pike estimator. A hazard ratio <1 indicates a lower risk with eltrombopag compared with Placebo. Log-rank test stratified by IVRS stratification factors; Test type: Superiority or Other; p = 0.164, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.97 to 2.08]

3. Secondary Outcome: Summary of Progression Free Survival From Investigator Assessment (ITT)
Description: Progression-free survival, defined as the time from randomization until either disease progression or death. The modified 2006 IWG criteria for MDS used for progression assessment For patients with: Less than 5% BM blasts: ≥ 50% increase in blasts to > 5% blasts; 5% - <10% BM blasts: ≥ 50% increase to > 10% blasts; 10% - <20% BM blasts: ≥ 50% increase to > 20% blasts; 20% - 30% BM blasts: ≥ 50% increase to > 30% blasts
Time Frame: First day of each cycle (Cycles 3+), at the end of therapy visit and every 3 months in follow-up for approximately 2 years
Population: The intent-to-treat (ITT) population included all the patients randomized in the study
Measure: Number; unit: participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 72 | 66
participants
  Death | 34 | 36
  Disease progression | 38 | 30

4. Secondary Outcome: Summary of Progression Free Survival From Central Review (ITT)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The intent-to-treat (ITT) population included all the patients randomized in the study
Measure: Number; unit: participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participants
  Death | 44 | 41
  Disease progression | 32 | 26

5. Secondary Outcome: Summary of AML Progression From Investigator Assessment and Central Review (ITT)
Description: Progression to AML in MDS patients with baseline bone marrow blast < 20% was defined as meeting definition of disease progression according to the modified 2006 IWG response criteria for MDS with the additional requirement that bone marrow blast or peripheral blast increases from < 20% at baseline to ≥ 20% postbaseline. Progression assessment For patients with:
  Less than 5% BM blasts: ≥ 50% increase in blasts to > 5% blasts; 5% - <10% BM blasts: ≥ 50% increase to > 10% blasts; 10% - <20% BM blasts: ≥ 50% increase to > 20% blasts; 20% - 30% BM blasts: ≥ 50% increase to > 30% blasts
Time Frame: as for outcome 3
Population: The intent-to-treat (ITT) population included all the patients randomized in the study
Measure: Number; unit: participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participants
  Participants progressed-AML - investigator assess | 27 | 16
  Participants progressed to AML - Central Review | 21 | 10

6. Secondary Outcome: Best Disease Response From Investigator Assessment (ITT)
Description: Best disease response is categorized as complete remission (CR), partial remission (PR), or marrow CR, stable disease, disease progression, or as non-evaluable; according to modified 2006 International Working Group (IWG) criteria for MDS
Time Frame: At end of Cycle 6 (cycle=28 days) or end of therapy, whichever came first
Measure: Number; unit: participant
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 140 | 150
participant
  Complete response - CR | 15 | 26
  Marrow complete response | 8 | 14
  Partial response - PR | 13 | 22
  Stable disease | 50 | 47
  Progressive disease | 22 | 8
  Not evaluable | 32 | 33
  Overall Response (CR+Marrow+PR | 36 | 62

7. Secondary Outcome: Best Disease Response From Central Review (ITT)
Description: as for outcome 6
Time Frame: At end of Cycle 6 (cycle=28 days) or end of therapy, whichever came first
Measure: Number; unit: participant
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 88 | 105
participant
  Complete response - CR | 11 | 7
  Marrow complete response | 2 | 5
  Partial response - PR | 2 | 7
  Stable disease | 23 | 31
  Progressive disease | 24 | 17
  Not evaluable | 26 | 38
  Overall Response (CR+Marrow+PR) | 15 | 19

8. Secondary Outcome: Hematologic Improvement (HI) in Platelets, Neutrophils, and Hemoglobin Based on the Modified IWG Criteria for MDS (ITT)
Description: HI based on the modified IWG criteria for MDS. HI - Platelets (BL <100Gi/L), response criteria= BL <20: increase to>20 and 100% at least for 56 days or BL >=20: absolute increase of >=30. HI - Neutrophils (BL <1.0 Gi/L), response criteria=100% increase and an absolute increase >0.5 Gi/L over BL for at least 56 days. HI-Hemoglobin (BL <g/dL), response criteria=Hgb increase by >=1.5 g/dL over BL, RBC transfusions(given for Hgb<=9.0) reduced by >=4 per 8w from BL
Time Frame: From Day 1 to 4-week follow-up (samples collected weekly in Cycle 1, Days 1 and 15 in Cycles 2-6 and Day 1 of Cycles >=7)
Measure: Number; unit: participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participants
  Platelets | 56 | 57
  Neutrophils | 12 | 13
  Hemoglobin | 1 | 1
  Platelets and neutrophils | 10 | 11
  Platelets and hemoglobin | 1 | 1
  Neutrophils and hemoglobin | 1 | 1
  Platelets, neutrophils and hemoglobin | 1 | 1

9. Secondary Outcome: Number of Participants Who Were Platelet Transfusion Independent (ITT Set)
Description: Platelet transfusion independence is defined for each cycle as the number of participants who continue to the end of a cycle without requiring a platelet transfusion
Time Frame: From Day 1 to end of study treatment up to approximately 2 years
Measure: Number; unit: participants
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participants
  Screening (179,177) | 127 | 121
  Cycle 1 (175,173) | 68 | 87
  Cycle 2 (135,158) | 62 | 87
  Cycle 3 (105,131) | 68 | 94
  Cycle 4 (93,116) | 58 | 91
  Cycle 5 (76,108) | 49 | 76
  Cycle 6 (65,90) | 41 | 62
  Cycle 7 (47,74) | 29 | 50
  Cycle 8 (37,61) | 20 | 42
  Cycle 9 (28,46) | 19 | 36
  Cycle 10 (23,38) | 18 | 28
  Cycle 11 (19,29) | 13 | 20
  Cycle 12 (15,21) | 10 | 15
  Cycle 13 (12,16) | 7 | 10
  Cycle 14 (6,11) | 3 | 6
  Cycle 15 (3,5) | 2 | 3
  Cycle 16 (0,3) | 0 | 3
  Cycle 17 (0,3) | 0 | 0

10. Secondary Outcome: Bleeding Adverse Events (AEs) >= Grade 3
Description: Bleeding will be assessed by recording AEs or serious adverse events (SAEs) as graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: From Day 1 to 4-week follow-up up to approximately 2 years
Measure: Number; unit: participant
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 177 | 177
participant
  Any event - Grade 3 | 9 | 12
  Any event - Grade 4 | 2 | 2
  Any event - Grade 5 | 1 | 4

11. Secondary Outcome: Number of of Subjects With Azacitidine Dose Delays, Dose Reductions, Interruptions
Description: The proportion of subjects with any delay, reduction or interruption in dosage of Azacitidine excluding those for non-medical reasons will be analyzed
Time Frame: From Day 1 to 4-week follow-up up to approximately 2 years
Measure: Number; unit: participant
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participant
  Overall dose delay | 82 | 88
  Overall dose reduction | 7 | 16
  Overall dose interruption | 3 | 13

12. Secondary Outcome: Response Levels in All Domains of Euroquol-5 Dimensions of Health, 3 Response Levels (EQ-5D-3L™)
Description: The EQ-5D is a general health status and health utility measure which captures 5 dimensions of health state: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. (EQ-5D is a trademark of the Stichting EuroQol Group) . C=cycle, D=Day
Time Frame: From Day 1 to 4-week follow-up up to approximately 2 years
Measure: Number; unit: participant
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
participant
  Mobility C1, D1 (176, 173) L1- no problem walking | 94 | 105
  Mobility C1,D1 (176, 173) L2- some problem walking | 81 | 66
  Mobility C1, D1 (176,173) L3- confined to bed | 1 | 2
  Mobility Wk 4 FU (71,72) L1- no problem walking | 40 | 48
  Mobility Wk 4 FU (71,72) L2- some problem walking | 29 | 22
  Mobility Wk 4 FU (71,72) L3- confined to bed | 2 | 2
  Self-Care C1, D1 (176,173) L1-no problems | 140 | 125
  Self-Care C1, D1 (176,173) L2-some problems | 32 | 20
  Self-Care C1, D1 (176,173) L3-unable to | 4 | 51
  Self-Care Wk4 FU (71,72) L1-no problems | 56 | 62
  Self-Care Wk4 FU(71,72) L2-some problems | 13 | 9
  Self-Care Wk4 FU (71,72) L2-unable to wash/dress | 2 | 1
  Usual activities C1,D1(175,173) L1-no problem | 97 | 94
  Usual activities C1,D1(175,173) L2-some problem | 71 | 68
  Usual activities C1,D1(175,173) L3-unable to | 7 | 11
  Usual activities Wk4 FU (71,72) L1-no problem | 36 | 41
  Usual activities Wk4 FU (71,72) L1-some problem | 29 | 25
  Usual activities Wk4 FU (71,72) L3-unable to | 6 | 6
  Pain/discomfort C1,D1(176,173) L1-none | 97 | 89
  Pain/discomfort C1,D1(176,173) L2-moderate | 74 | 78
  Pain/discomfort C1,D1(176,173) L3-extreme | 5 | 6
  Pain/discomfort Wk4 FU (71,72) L1-none | 38 | 40
  Pain/discomfort Wk4 FU (71,72) L2-moderate | 28 | 27
  Pain/discomfort Wk4 FU (71,72) L3-extreme | 5 | 5
  Anxiety/depression C1 D1(176,173) L1-none | 96 | 112
  Anxiety/depression C1 D1(176,173) L2-moderately | 74 | 56
  Anxiety/depression C1 D1(176,173) L3-extremely | 6 | 5
  Anxiety/depression Wk4 FU(71,72) L1-none | 44 | 45
  Anxiety/depression Wk4 FU(71,72) L2-moderately | 24 | 25
  Anxiety/depression Wk4 FU(71,72) L3-extremely | 3 | 2

13. Secondary Outcome: Functional Assessment of Chronic Disease Therapy-fatigue Subscale (FACIT-Fatigue) (ITT)
Description: The FACIT-Fatigue subscale measures severity and impact of fatigue on functioning and Health Related QoL experienced in the past 7 days. Scale is a 13 item measure of fatigure. Items are scored on a 0-4 response scale ranging from "not at all" to "very much so". All items are summed to create a single fatigure score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatiigue (The FACIT Fatigue Scale is owned by David Cella, Ph.D.)
Time Frame: From Day 1 to 4-week follow-up (Approximate median 9 Cycles+4 weeks follow-up) up to approximately 2 years
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
scores
  Cycle 1 Day 1 (175,172) | 17.401 (11.0279) | 15.951 (10.9911)
  Week 4 Follow-up (68,70) | 16.669 (10.7266) | 14.898 (12.2362)

14. Secondary Outcome: Medical Resource Utilization (MRU): Event -Hospitalizations Inpatient and Outpatient
Description: MRU data will be collected for each subject. Events corresponding to unscheduled (not scheduled per protocol) hospitalizations
Time Frame: From Day 1 to 4-week follow-up (Approximate median 9 Cycles+4 weeks follow-up) up to approximately 2 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
days
  In-patient hospitalizations - entire study (91,66) | 23.9 (24.33) | 27.1 (33.81)
  Out-patient hospitalizations - entire study (4,2) | 9.5 (16.34) | 2.5 (0.71)

15. Secondary Outcome: Medical Resource Utilization (MRU): Event and Use of Site Specific Medical Resources - Non-study Laboratory Tests
Description: MRU data will be collected for each subject. Events corresponding to unscheduled (not scheduled per protocol) hospitalizations, office visits including consultations, laboratory and diagnostic tests (lab results, imaging etc.), and procedures prior to therapy initiation and during therapy will be collected
Time Frame: From Day 1 to 4-week follow-up (Approximate median 9 Cycles+4 weeks follow-up) up to approximately 2 years
Measure: Number; unit: tests
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
tests | 88 | 105

16. Secondary Outcome: Medical Resource Utilization (MRU): Use of Site Specific Medical Resources
Description: as for outcome 15
Time Frame: From Day 1 to 4-week follow-up (Approximate median 9 Cycles+4 weeks follow-up) up to approximately 2 years
Measure: Number; unit: visits
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 179 | 177
visits
  Medical or surgical specialist visits | 49 | 58
  Home healthcare visits by medical professional | 89 | 97
  Primary physician care visits | 89 | 97
  Nurse practitioner, physic assistant, nurse visits | 89 | 97
  Telephone consultations | 89 | 97
  Emergency visits not resulting in hospital stay | 89 | 97

17. Secondary Outcome: Summary of Post-Hoc Estimates of Steady-state Eltrombopag Cmax and Cmin Pharmacokinetic Parameters for a 50 mg Dose
Description: Eltrombopag concentrations were analyzed using a population PK model along with data from other studies in healthy volunteers and in patients with MDS and/or AML. Post-hoc PK parameters were derived. Only patients from this study were included (163)
Time Frame: Cycle 1, Week 2: Pre-dose, 1.5 and 3 hour post dose; Cycle 1, Week 3: 4, 5.5, and 7 hours post dose
Population: All patients with evaluable eltrombopag dosing, actual sampling time, and eltrombopag concentration data were included in the population PK dataset and analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 163
μg/mL
  Cmax | 7.70 (36.8)
  Cmin | 4.41 (49.9)

18. Secondary Outcome: Summary of Post-Hoc Estimates of Steady-state Eltrombopag AUC0 Infinity Pharmacokinetic Parameters for a 50 mg Dose
Description: as for outcome 17
Time Frame: Cycle 1, Week 2: Pre-dose, 1.5 and 3 hour post dose; Cycle 1, Week 3: 4, 5.5, and 7 hours post dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.μg/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 163
hr.μg/mL | 135 (43.1)

19. Secondary Outcome: AUC0-infinity -Pharmacokinetic(s) Parameter of Azacitidine
Description: An analysis of variance (ANOVA) on AUC0-infinity. The PK parameters were log transformed prior to analysis. The model included treatment as a fixed effect. Point estimates and their associated 90% CI were constructed for the differences in PK parameter values. The point estimates and their associated 90% CI were then back transformed to provide point estimates and 90% CI for the azacitidine + eltrombopag:azacitidine + placebo PK parameter ratios.
Time Frame: Cycle 2 Day 1: Pre-dose, 15 min, 0.5, 1, 2 and 4 hr post dose
Population: all patients with evaluable azacitidine dosing, actual sampling time, and azacitidine concentration data were included in the NCA dataset and analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.ng/mL
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 22 | 23
hr.ng/mL | 840 (53) | 641 (67)
Statistical Analysis 1: Comparison: Eltrombopag vs Placebo; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 1.31, 90% CI 2-sided [0.990 to 1.74]

20. Secondary Outcome: Cmax -Pharmacokinetic Parameter of Azacitidine
Description: An analysis of variance (ANOVA) on Cmax . The PK parameters were log transformed prior to analysis. The model included treatment as a fixed effect. Point estimates and their associated 90% CI were constructed for the differences in PK parameter values. The point estimates and their associated 90% CI were then back transformed to provide point estimates and 90% CI for the azacitidine + ltrombopag:azacitidine + placebo PK parameter ratios.
Time Frame: Cycle 2 Day 1: Pre-dose, 15 min, 0.5, 1, 2 and 4 hr post dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Eltrombopag | Placebo
Number analyzed (Participants) | 26 | 26
ng/mL | 744 (91) | 535 (89)
Statistical Analysis 1: Comparison: Eltrombopag vs Placebo; Test type: Superiority or Other; ANOVA; Geometric mean ratio = 1.39, 90% CI 2-sided [0.970 to 1.99]

ADVERSE EVENTS:
Time Frame: Timeframe for AE
Description: AE additional description
Groups:
- Eltrombopag: Eltrombopag
- Placebo: Placebo
Arm/Group | Eltrombopag | Placebo
Serious Adverse Events (participants affected / at risk) | 128/177 | 100/177
Other Adverse Events (participants affected / at risk) | 159/177 | 153/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=177) | Placebo (N=177)
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Cytopenia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 47 | 33
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardiovascular deconditioning (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Papillary muscle infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 5
Gingival bleeding (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 2
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 3 | 3
Inflammation (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Mucosal haemorrhage (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 20 | 8
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 2
Anal abscess (Infections and infestations) | 1 | 0
Anal fistula infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 1
Carbuncle (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 6 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 2
Extradural abscess (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1
Fungal pharyngitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 4
Infectious colitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 20 | 17
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyomyositis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 10 | 7
Septic shock (Infections and infestations) | 10 | 5
Skin infection (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 1
Tongue fungal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 5
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood osmolarity decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 2
Haematuria (Renal and urinary disorders) | 0 | 3
Nephritis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic dilatation (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=177) | Placebo (N=177)
Anaemia (Blood and lymphatic system disorders) | 32 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 10
Leukopenia (Blood and lymphatic system disorders) | 9 | 5
Neutropenia (Blood and lymphatic system disorders) | 52 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 14
Abdominal pain (Gastrointestinal disorders) | 7 | 12
Abdominal pain upper (Gastrointestinal disorders) | 9 | 7
Constipation (Gastrointestinal disorders) | 48 | 57
Diarrhoea (Gastrointestinal disorders) | 42 | 25
Gingival bleeding (Gastrointestinal disorders) | 13 | 9
Nausea (Gastrointestinal disorders) | 54 | 46
Stomatitis (Gastrointestinal disorders) | 9 | 3
Vomiting (Gastrointestinal disorders) | 33 | 29
Asthenia (General disorders) | 28 | 34
Chills (General disorders) | 8 | 11
Fatigue (General disorders) | 31 | 27
Injection site pain (General disorders) | 7 | 9
Oedema peripheral (General disorders) | 22 | 11
Pyrexia (General disorders) | 44 | 40
Nasopharyngitis (Infections and infestations) | 7 | 9
Pneumonia (Infections and infestations) | 12 | 9
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Urinary tract infection (Infections and infestations) | 9 | 8
Alanine aminotransferase increased (Investigations) | 10 | 3
Blood bilirubin increased (Investigations) | 13 | 2
Neutrophil count decreased (Investigations) | 12 | 11
Platelet count decreased (Investigations) | 9 | 5
White blood cell count decreased (Investigations) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 27 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 14
Dizziness (Nervous system disorders) | 17 | 14
Headache (Nervous system disorders) | 20 | 13
Insomnia (Psychiatric disorders) | 16 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 18
Erythema (Skin and subcutaneous tissue disorders) | 11 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 11 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 12
Rash (Skin and subcutaneous tissue disorders) | 19 | 11
Haematoma (Vascular disorders) | 10 | 12
Hypertension (Vascular disorders) | 2 | 11
Hypotension (Vascular disorders) | 12 | 5

LIMITATIONS AND CAVEATS:
The IDMC recommended terminating the study for futility (primary) and safety (secondary). Due to early termination of the trial, the final analysis of OS took place at the same time as the final analysis of the primary end point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novaratis does not prohibit any investigation from publishing. Any publications from a single-site are postposed until the publication of the pooled data (ie. data from all sites) in the clinical trial.